CLINICAL TRIAL: NCT02453386
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Determine the Efficacy and Safety of Tozadenant as Adjunctive Therapy in Levodopa-Treated Patients With Parkinson's Disease Experiencing End of Dose "Wearing-Off" (TOZ-PD)
Brief Title: Safety and Efficacy Study of Tozadenant to Treat End of Dose Wearing Off in Parkinson's Patients
Acronym: TOZ-PD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: New Safety Information
Sponsor: Biotie Therapies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TOZ-CL05; 2014-005630-60 (EudraCT Number)
Record Dates: First submitted 2015-05-21; First posted 2015-05-25 (Estimated); Results first posted 2019-03-26 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-03

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Motor fluctuations; Off time; On time; Dyskinesia
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — tozadenant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tozadenant 60 mg BID (Experimental): During Part A, patients took two (2) tablets, one 60 mg tozadenant and one placebo, by mouth BID for a total of four (4) tablets per day.
  Upon completion of Part A, all patients will begin dosing with open label tozadenant in Part B.
  Interventions: Drug: tozadenant
- Tozadenant 120 mg BID (Experimental): During Part A, patients took two (2) tablets of 60 mg tozadenant, by mouth BID for a total of four (4) tablets per day.
  Upon completion of Part A, all patients will begin dosing with open label tozadenant in Part B.
  Interventions: Drug: tozadenant
- Placebo BID (Placebo Comparator): During Part A, patients took two (2) tablets of placebo, by mouth BID for a total of four (4) tablets per day.
  Upon completion of Part A, all patients will begin dosing with open label tozadenant in Part B.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: tozadenant
  Other Names: SYN115
  Arms: Tozadenant 120 mg BID; Tozadenant 60 mg BID
Drug: placebo
  Other Names: tozadenant placebo
  Arms: Placebo BID

SUMMARY:
Phase 3, international, multicenter, randomized, double-blind, placebo-controlled, parallel-group, 3-arm safety and efficacy study (Part A) with an open-label phase (Part B).

DETAILED DESCRIPTION:
During Part A, each patient will participate for up to 30 weeks, which includes a Screening Period of 1 to ≤ 6 weeks, followed by a Baseline Visit and 24 weeks of double-blind treatment:

* Screening Period: 1 - 6 weeks.
* Double-Blind Treatment Period: 24 weeks.

After completion of Part A, patients will continue in Part B for an additional 56 weeks:

* Open-Label Treatment Period: 52 weeks.
* Post-Treatment Safety Follow Up: 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient understands study requirements and has given his/her written informed consent on an Institutional Review Board (IRB) or Independent Ethics Committee (IEC) approved consent form.
* Parkinson's disease diagnosis consistent with UK Parkinson's Disease Society Brain Bank Diagnostic criteria
* Minimum of 3 years since diagnosis.
* Meet Hoehn and Yahr PD stage
* Good response to levodopa
* Stable regimen of anti-PD medications
* Patients must have been taking a levodopa-containing anti-PD medication continuously for at least the previous 12 months
* Patient has documented a minimum amount of Off time.
* If of childbearing potential (male and female) must use an acceptable method of contraception

Exclusion Criteria:

* Previous tozadenant study participation
* Current or recent participation in another study.
* Secondary or atypical parkinsonism
* Neurosurgical intervention for PD
* Patient is taking apomorphine, budipine, istradefylline, tolcapone, or DUOPA™/Duodopa®
* Treatment with excluded medications
* Untreated or uncontrolled hyperthyroidism or hypothyroidism
* Clinically significant out-of-range laboratory
* MMSE out of range
* Current episode of major depression (stable treatment for depression is permitted).
* Recent suicide attempt or suicidal ideation type 4 or type 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS)
* Women lactating or pregnant
* Hypersensitivity to any components of tozadenant or excipients
* Abnormal findings on the physical or neurological examination, or medical history that would make the patient unsuitable for the study
* History of hepatitis or cholangitis

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2018-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Kenney, MD, Study Director — Biotie Inc.
Locations (71):
- United States (40):
  - Birmingham, Alabama
  - Sun City, Arizona
  - Loma Linda, California
  - Los Angeles, California
  - Oxnard, California
  - Reseda, California
  - Sacramento, California
  - Sunnyvale, California
  - Englewood, Colorado
  - Vernon, Connecticut
  - Boca Raton, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Chicago, Illinois
  - Kansas City, Kansas
  - Lexington, Kentucky
  - Baltimore, Maryland
  - Boston, Massachusetts
  - East Lansing, Michigan
  - Farmington Hills, Michigan
  - West Bloomfield, Michigan
  - St Louis, Missouri
  - Albany, New York
  - Commack, New York
  - Rochester, New York
  - Asheville, North Carolina
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Toledo, Ohio
  - Tulsa, Oklahoma
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Houston, Texas
  - Burlington, Vermont
  - Roanoke, Virginia
  - Kirkland, Washington
- Austria (2):
  - Innsbruck
  - Vienna
- Canada (3):
  - Edmonton, Alberta
  - Ottawa, Ontario
  - Toronto, Ontario
- Czechia (5):
  - Brno
  - Choceň
  - Pardubice
  - Prague
  - Rychnov nad Kněžnou
- Germany (6):
  - Beelitz-Heilstätten
  - Berlin
  - Dresden
  - Haag in Oberbayern
  - Marburg
  - Ulm
- Italy (9):
  - Arcugnano
  - Cassino
  - Chieti
  - Grosseto
  - Pavia
  - Pisa
  - Rome
  - Salerno
  - Venice
- Spain (6):
  - Manresa, Barcelona
  - Sant Cugat del Vallès, Barcelona
  - Terrassa, Barcelona
  - Donostia / San Sebastian, Guipuzcoa
  - Barcelona
  - Madrid

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 80 sites in 7 countries. Planned patient enrollment numbers were achieved, but the study and the tozadenant development program were terminated prior to study completion by all patients, based on an unexpected emerging safety signal as discussed in the safety sections of this report.
Groups:
- Tozadenant 60 mg BID: During Part A, patients took two (2) tablets, one 60 mg tozadenant and one placebo, by mouth BID for a total of four (4) tablets per day.
- Tozadenant 120 mg BID: During Part A, patients took two (2) tablets of 60 mg tozadenant, by mouth BID for a total of four (4) tablets per day.
- Placebo BID: During Part A, patients took two (2) tablets of placebo, by mouth BID for a total of four (4) tablets per day.
Period: Overall Study
Arm/Group | Tozadenant 60 mg BID | Tozadenant 120 mg BID | Placebo BID
Started | 151 | 149 | 149
Completed | 102 | 100 | 108
Not Completed | 49 | 49 | 41
Not completed — Adverse Event | 22 | 30 | 15
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Withdrawal by Subject | 10 | 9 | 9
Not completed — Sponsor Terminated Study | 14 | 8 | 11
Not completed — Subject Terminated by Sponsor | 1 | 1 | 1
Not completed — Sponsor Terminated by Investigator | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Other | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The 449 patients who were randomized in the study comprised the ITT set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tozadenant 60 mg BID | Tozadenant 120 mg BID | Placebo BID | Total
Number analyzed (Participants) | 151 | 149 | 149 | 449
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 73 | 61 | 66 | 200
  >=65 years | 78 | 88 | 83 | 249
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (8.68) | 65.1 (7.57) | 65.0 (8.29) | 64.7 (8.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 49 | 48 | 148
  Male | 100 | 100 | 101 | 301
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 5 | 15
  Not Hispanic or Latino | 146 | 144 | 144 | 434
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 2 | 2 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 2
  White | 148 | 144 | 146 | 438
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 5 | 5 | 5 | 15
  Austria | 3 | 3 | 2 | 8
  United States | 69 | 69 | 69 | 207
  Czechia | 22 | 22 | 22 | 66
  Italy | 20 | 19 | 20 | 59
  Germany | 19 | 19 | 19 | 57
  Spain | 13 | 12 | 12 | 37
Weight at Screening [Mean (Standard Deviation); unit: kilograms] | 78.74 (15.725) | 80.42 (16.576) | 79.35 (14.436) | 79.50 (15.585)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 24 in the Number of Hours Per Day Spent in OFF Time
Description: Awake time in OFF state (hr) is the average of maximum of 3 days diary. The primary efficacy endpoint was the change from baseline to Week 24 in OFF time, where OFF time in the Hauser Parkinson's Disease Home Diary (PD) was averaged over 3 days prior to the study visit. During Screening and through Part A of the study, the Hauser Parkinson's Disease Home Diary (PD) was completed on specified days directly preceding the scheduled study visits/assessments. Motor activity was recorded as OFF, ON (mobility improved), or asleep time. Patients were asked to record ON time according to dyskinesia categories "without dyskinesia", "with non troublesome dyskinesia" or "with troublesome dyskinesia". Patients (and/or caregivers) were trained to complete the PD diary to record their status at half hourly intervals as OFF, ON without dyskinesia, ON with non troublesome dyskinesia, ON with troublesome dyskinesia, or asleep.
Time Frame: Baseline to 24 Weeks
Population: Modified Intent-to-Treat (mITT) population
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Placebo BID: Two placebo tablets BID
- Tozadenant 60 mg BID: One 60 mg tozadenant tablet BID plus 1 Placebo
- Tozadenant 120 mg BID: Two 60 mg tozadenant tablets BID
Arm/Group | Placebo BID | Tozadenant 60 mg BID | Tozadenant 120 mg BID
Number analyzed (Participants) | 145 | 144 | 145
hours
  Baseline | 6.34 (1.986) | 6.00 (1.970) | 6.25 (2.337)
  Week 2: number analyzed (Participants) | 145 | 143 | 145
  Week 2 | -0.725 (2.0018) | -1.100 (2.1188) | -1.409 (2.3957)
  Week 6: number analyzed (Participants) | 139 | 139 | 134
  Week 6 | -0.817 (2.0993) | -1.112 (2.2903) | -1.879 (2.2866)
  Week 12: number analyzed (Participants) | 130 | 128 | 122
  Week 12 | -0.962 (2.2186) | -1.460 (2.3689) | -1.919 (2.2008)
  Week 18: number analyzed (Participants) | 119 | 117 | 113
  Week 18 | 0.860 (2.4246) | -1.020 (2.5886) | -1.742 (2.6855)
  Week 24: number analyzed (Participants) | 108 | 104 | 104
  Week 24 | -0.958 (2.2725) | -0.835 (2.9730) | -1.789 (2.4802)

2. Secondary Outcome: Change in Good ON Time From Baseline to Week 24
Description: The first key secondary efficacy endpoint was the change from baseline to Week 24 in good ON which was defined as ON without dyskinesia or ON with non-troublesome dyskinesia.
  Awake Time in Good ON State (hr) is the average of a maximum of 3 days diary. Patients were asked to record ON time according to dyskinesia categories "without dyskinesia", "with non troublesome dyskinesia" or "with troublesome dyskinesia" . Patients (and/or caregivers) were trained to complete the PD diary to record their status at half hourly intervals as OFF, ON without dyskinesia, ON with non troublesome dyskinesia, ON with troublesome dyskinesia, or asleep. For patients with missing baseline or baseline was measured post-dose, screening was used as baseline in the calculation of change from baseline.
Time Frame: Baseline to 24 Weeks
Population: Modified Intent-to-Treat (mITT) population
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Placebo: One placebo BID
- 120 mg Tozadanent: Two 60 mg tozadenant tablets BID
Arm/Group | Placebo | Tozadenant 60 mg BID | 120 mg Tozadanent
Number analyzed (Participants) | 145 | 144 | 145
hours
  Baseline | 9.58 (2.266) | 9.92 (2.217) | 9.51 (2.554)
  Week 2: number analyzed (Participants) | 145 | 143 | 145
  Week 2 | 0.790 (2.2778) | 1.145 (2.1291) | 1.397 (2.5102)
  Week 6: number analyzed (Participants) | 139 | 139 | 134
  Week 6 | 0.812 (2.4177) | 1.002 (2.4533) | 1.650 (2.2538)
  Week 12: number analyzed (Participants) | 130 | 128 | 122
  Week 12 | 0.777 (2.4300) | 1.307 (2.7051) | 1.830 (2.2870)
  Week 18: number analyzed (Participants) | 119 | 117 | 113
  Week 18 | 0.709 (2.6284) | 0.903 (2.6297) | 1.553 (2.6138)
  Week 24: number analyzed (Participants) | 108 | 104 | 104
  Week 24 | 1.011 (2.5470) | 0.705 (3.1219) | 1.689 (2.7335)

3. Secondary Outcome: Change in Unified Parkinson's Disease Rating Scale (UPDRS) Part II Activities of Daily Living (ADL) Subscale + Part III Motor Function
Description: The Unified Parkinson's Disease Rating Scale (UPDRS) is a scale to monitor Parkinson's Disease related disability and impairment. The scale itself has 4 components are titled; (1) nonmotor experiences of daily living (13 items), (2) motor experiences of daily living (13 items), (3) motor examination (18 items), and (4) motor complications (six items). Each subscale now has 0-4 ratings, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. In this outcome measure we are evaluating Part II and Part III.
  Part II: self-evaluation of the activities of daily life (ADLs) including speech, swallowing, handwriting, dressing, hygiene, falling, salivating, turning in bed, walking, and cutting food Part III: clinician-scored monitored motor evaluation Range of score is 0 - 160: 0 meaning less impact and Higher score indicates greater impact of PD symptoms.
Time Frame: Baseline to Week 24
Population: mITT population (Modified Intent-to-Treat) - all safety set patients who had valid diaries at baseline and had valid diaries on at least 1 post-baseline visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Tozadenant 60 mg: One 60 mg tozadenant tablet BID plus 1 Placebo
- Tozadenant 120 mg: Two 60 mg tozadenant tablets BID
Arm/Group | Placebo | Tozadenant 60 mg | Tozadenant 120 mg
Number analyzed (Participants) | 145 | 144 | 145
score on a scale
  Baseline: number analyzed (Participants) | 140 | 141 | 143
  Baseline | 33.2 (12.14) | 31.3 (12.18) | 32.3 (12.08)
  Week 2: number analyzed (Participants) | 143 | 141 | 142
  Week 2 | -3.16 (5.931) | -3.43 (6.611) | -3.96 (5.924)
  Week 6: number analyzed (Participants) | 136 | 138 | 131
  Week 6 | -3.53 (6.375) | -2.82 (7.223) | -4.31 (6.362)
  Week 12: number analyzed (Participants) | 130 | 127 | 118
  Week 12 | -3.02 (8.385) | -3.64 (7.393) | -4.38 (6.602)
  Week 18: number analyzed (Participants) | 118 | 113 | 111
  Week 18 | -3.35 (7.934) | -3.63 (7.958) | -3.83 (7.150)
  Week 24: number analyzed (Participants) | 108 | 103 | 106
  Week 24 | -2.80 (8.183) | -2.54 (8.584) | -3.68 (7.853)

4. Secondary Outcome: Change From Baseline to Week 24 in the ON State in Unified Parkinson's Disease Rating Scale (UPDRS) Part IIl
Description: Change from Baseline to Week 24 in the Unified Parkinson's Disease Rating Scale (UPDRS) Parts III Motor Function (motor subscale) total scores. Each subscale has 0-4 ratings, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. Range of score is 0 - 108. Higher scores indicate greater impact of PD symptoms. Unified Parkinson's Disease Rating Scale (UPDRS) in the ON state was measured at a time representative of the ON state in that patient, not in "best" ON. Unified Parkinson's Disease Rating Scale Part III in OFF was not evaluated.
Time Frame: Baseline to Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Tozadenant 60 mg | Tozadenant 120 mg
Number analyzed (Participants) | 145 | 144 | 145
score on a scale
  Baseline: number analyzed (Participants) | 140 | 141 | 143
  Baseline | 20.9 (8.80) | 19.8 (8.58) | 20.5 (8.71)
  Week 2: number analyzed (Participants) | 143 | 141 | 142
  Week 2 | -2.13 (4.828) | -2.35 (5.144) | -2.83 (4.613)
  Week 6: number analyzed (Participants) | 136 | 138 | 131
  Week 6 | -2.29 (5.011) | -2.18 (5.476) | -2.76 (5.423)
  Week 12: number analyzed (Participants) | 130 | 127 | 118
  Week 12 | -2.31 (6.276) | -2.69 (5.822) | -3.19 (5.356)
  Week 18: number analyzed (Participants) | 118 | 113 | 111
  Week 18 | -2.46 (6.112) | -2.64 (6.303) | -2.95 (5.572)
  Week 24: number analyzed (Participants) | 108 | 103 | 106
  Week 24 | -2.15 (6.363) | -2.13 (6.822) | -2.93 (6.048)

5. Other Pre Specified Outcome: Global Assessments of Improvement: Clinical Global Impression of Improvement (CGI-I) Week 24
Description: For the Clinical Global Impression of Improvement (CGI-I), the investigator or rater is asked to rate the patient's total improvement, whether or not in his or her judgment it is due entirely to drug treatment, based on a 1-7 point weighted scale ranging from "very much improved" (1) to "very much worse" (7). A zero score is assigned if the score is not assessed. Scale: 1 = Very much improved, 2 = Much improved, 3 = Minimally improved, 4 = No change, 5 = Minimally worse, 6 = Much worse, 7 = Very much worse. Tables show Treatment vs Placebo.
Time Frame: At Week 24
Population: mITT population (Modified Intent-to-Treat) - all safety set patients who had valid diaries at baseline and had valid diaries on at least 1 post-baseline visit. Patients were accounted for in the treatment group to which they were originally randomized.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: One Placebo
- Tozadanent 120 mg: Two 60 mg tozadenant tablets BID
Arm/Group | Placebo | Tozadenant 60 mg | Tozadanent 120 mg
Number analyzed (Participants) | 145 | 144 | 145
score on a scale
  Week 2: number analyzed (Participants) | 145 | 144 | 144
  Week 2 | 3.5 (0.80) | 3.4 (0.87) | 3.2 (0.85)
  Week 6: number analyzed (Participants) | 138 | 138 | 133
  Week 6 | 3.4 (0.86) | 3.3 (0.96) | 3.2 (0.93)
  Week 12: number analyzed (Participants) | 132 | 129 | 122
  Week 12 | 3.5 (0.98) | 3.3 (1.01) | 3.2 (0.92)
  Week 18: number analyzed (Participants) | 120 | 117 | 114
  Week 18 | 3.5 (1.04) | 3.5 (0.92) | 3.2 (0.97)
  Week 24: number analyzed (Participants) | 111 | 106 | 107
  Week 24 | 3.5 (0.92) | 3.5 (1.07) | 3.2 (0.98)

6. Other Pre Specified Outcome: Patient Global Impression of Improvement (PGI-I) Week 24
Description: For the Patient Global Impression of Improvement (PG-I), the patient is asked to rate the total improvement of their Parkinson's Disease, whether or not in the patient's judgment it is due entirely to drug treatment, based on a 1-7 point weighted scale. "very much improved" (1) to "very much worse" (7). A zero score is assigned if the score is not assessed.
  Scale: 1 = Normal, not at all ill, 2 = Borderline ill, 3 = Mildly ill, 4 = Moderately ill, 5 = Markedly ill, 6 = Severly ill, 7 = Among the most extremely ill.
  Tables show Treatment vs Placebo.
Time Frame: At Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Tozadenant 60 mg | Tozadenant 120 mg
Number analyzed (Participants) | 145 | 144 | 145
score on a scale
  Week 2: number analyzed (Participants) | 145 | 144 | 144
  Week 2 | 3.6 (0.90) | 3.3 (1.02) | 3.1 (1.00)
  Week 6: number analyzed (Participants) | 138 | 140 | 134
  Week 6 | 3.5 (0.92) | 3.4 (1.22) | 3.1 (1.02)
  Week 12: number analyzed (Participants) | 132 | 129 | 122
  Week 12 | 3.5 (1.16) | 3.5 (1.21) | 3.1 (1.13)
  Week 18: number analyzed (Participants) | 120 | 117 | 114
  Week 18 | 3.6 (1.03) | 3.6 (1.13) | 3.2 (1.08)
  Week 24: number analyzed (Participants) | 111 | 106 | 107
  Week 24 | 3.6 (1.14) | 3.6 (1.21) | 3.4 (1.14)

ADVERSE EVENTS:
Time Frame: 24 Weeks
Description: The Adverse Events was based on the Safety Set Population (SS). The SS included 447 of the 449 (ITT Population) randomized patients as two patients who were randomized were not dosed.
Groups:
- Tozadenant 60 mg BID: Part A (double-blind phase)
  During Part A, patients took two (2) tablets, one 60 mg tozadenant and one placebo, by mouth BID for a total of four (4) tablets per day.
- Tozadenant 120 mg BID: Part A (double-blind phase)
  During Part A, patients took two (2) tablets of 60 mg tozadenant, by mouth BID for a total of four (4) tablets per day.
- Placebo BID: Part A (double-blind phase)
  During Part A, patients took two (2) tablets of placebo, by mouth BID for a total of four (4) tablets per day.
Arm/Group | Tozadenant 60 mg BID | Tozadenant 120 mg BID | Placebo BID
All-Cause Mortality (participants affected / at risk) | 1/150 | 1/149 | 1/148
Serious Adverse Events (participants affected / at risk) | 13/150 | 12/149 | 15/148
Other Adverse Events (participants affected / at risk) | 115/150 | 111/149 | 111/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tozadenant 60 mg BID (N=150) | Tozadenant 120 mg BID (N=149) | Placebo BID (N=148)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Torsade de pointes (Cardiac disorders) | 0 | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Burns third degree (Injury, poisoning and procedural complications) | 0 | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0
Carotid artery occlusion (Nervous system disorders) | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Dyskinesia (Nervous system disorders) | 1 | 0 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 1
Parkinson's disease (Nervous system disorders) | 2 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 2 | 0
Anuria (Renal and urinary disorders) | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0
Accelerated hypertension (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tozadenant 60 mg BID (N=150) | Tozadenant 120 mg BID (N=149) | Placebo BID (N=148)
Constipation (Gastrointestinal disorders) | 15 | 8 | 2
Dry Mouth (Gastrointestinal disorders) | 2 | 4 | 0
Nausea (Gastrointestinal disorders) | 8 | 13 | 6
Fatigue (General disorders) | 7 | 4 | 2
Nasopharyngitis (Infections and infestations) | 7 | 5 | 10
Urinary Tract Infection (Infections and infestations) | 4 | 9 | 4
Contusion (Injury, poisoning and procedural complications) | 0 | 5 | 1
Fall (Injury, poisoning and procedural complications) | 22 | 13 | 9
Blood creatine phosphokinase increased (Investigations) | 4 | 6 | 3
Weight decreased (Investigations) | 4 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 7 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 3 | 6
Dizziness (Nervous system disorders) | 7 | 7 | 9
Somnolence (Nervous system disorders) | 5 | 8 | 5
Sudden onset of sleep (Nervous system disorders) | 7 | 7 | 4
Anxiety (Psychiatric disorders) | 5 | 2 | 3
Hallucination, visual (Psychiatric disorders) | 8 | 8 | 2
Insomnia (Psychiatric disorders) | 9 | 9 | 9
Micturition urgency (Renal and urinary disorders) | 3 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 2
Flushing (Vascular disorders) | 1 | 4 | 1
Dyskinesia (Nervous system disorders) | 22 | 22 | 13
Confusional state (Psychiatric disorders) | 2 | 4 | 1
Parkinson's disease (Nervous system disorders) | 11 | 3 | 7
Upper respiratory tract infection (Infections and infestations) | 6 | 1 | 7
Hypertension (Vascular disorders) | 5 | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 6
White Blood cell count decreased (Investigations) | 2 | 0 | 4
Headache (Nervous system disorders) | 3 | 2 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1
Disorientation (Psychiatric disorders) | 4 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding the study results for a period up to 30 days from the date the communication is submitted to the sponsor. The sponsor shall have the right to defer proposed publication an additional 60 days from the end of the review period. The sponsor cannot require changes to the communication and cannot unilaterally extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-10-13): https://cdn.clinicaltrials.gov/large-docs/86/NCT02453386/Prot_000.pdf
  • Statistical Analysis Plan (2015-05-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT02453386/SAP_001.pdf